CLINICAL TRIAL: NCT06290310
Title: Assessment of Patient-ventilator Asynchrony by Electric Impedance Tomography and Artificial Intelligence
Brief Title: Assessment of Patient-ventilator Asynchrony by Electric Impedance Tomography
Acronym: PAVELA
Status: Not yet recruiting | Type: Observational
Sponsor: Kiskunhalas Semmelweis Hospital the Teaching Hospital of the University of Szeged (Other Government)
Collaborators: Hochschule Furtwangen University (Other); Budapest University of Technology and Economics (Other); Szeged University (Other)
Responsible Party: Sponsor
Other Study IDs: PAVELA
Record Dates: First submitted 2024-02-09; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Acute Lung Injury
Keywords: artificial intelligence; biotrauma; electric impedance tomography; patient-ventilator asynchrony
MeSH Terms: conditions — Acute Lung Injury; Patient-Ventilator Asynchrony

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mechanically ventilated patients: Invasively or non-invasively ventilated patients.
  Interventions: Device: EIT; Device: patient-ventilator asynchrony assessment

INTERVENTIONS:
Device: EIT — continuous electric impedance tomography measurement
Device: patient-ventilator asynchrony assessment — patient-ventilator asynchrony assessment by flow/time curve and machine learning

SUMMARY:
Patient-ventilator asynchrony (PVA) has deleterious effects on the lungs. PVA can lead to acute lung injury and worsening hypoxemia through biotrauma. Little is known about how PVA affects lung aeration estimated by electric impedance tomography (EIT). Artificial intelligence can promote the detection of PVA and with its help, EIT measurements can be correlated to asynchrony.

DETAILED DESCRIPTION:
Patient-ventilator asynchrony (PVA) is a common phenomenon with invasively- and non-invasively ventilated patients. PVA has deleterious effects on the lungs. It causes not just patient discomfort and distress but also leads to acute lung injury and worsening hypoxemia through biotrauma. The latter significantly impacts outcomes and increases the duration of mechanical ventilation and intensive care unit stay.

However, PVA is a widely investigated incident related to mechanical ventilation, though little is known about how it affects lung aeration estimated by electric impedance tomography (EIT). EIT is a non-invasive, real-time monitoring technique suitable for detecting changes in lung volumes during ventilation.

Artificial intelligence can promote the detection of PVA by flow versus time assessment. If continuous EIT recording is correlated with the latter, impedance tomography changes evoked by asynchrony can be estimated

ELIGIBILITY:
Inclusion Criteria:

* any patient ventilated invasively
* any patient ventilated non-invasively

Exclusion Criteria:

* age under 18

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: mechanically ventilated patients
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-04-12 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
distribution | during mechanical ventilation
  gas distribution in lungs assessed by electric impedance tomography

SECONDARY OUTCOMES:
connecting asysnchrony cycles with electric impedance tomography measurements | during mechanical ventilation
  connecting machine learning assessed patient-ventilator asynchrony respiratory cycles with the inherent respiratory cycle recorded by the electric impedance tomography
identifying unic electric impedance tomography signs of asynchrony | during mechanical ventilation
  following connection described under "outcome 2", identification if single patient-ventilator asynchrony types (delayed cycling, premature cycling, auto trigger, ineffective effort, double trigger) present specific electric impedance tomography changes

CONTACTS AND LOCATIONS:
Locations (1):
- Kiskunhalas Semmelweis Hopsital the Teaching Hospital of the University of Szeged, Kiskunhalas, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sottile PD, Albers D, Smith BJ, Moss MM. Ventilator dyssynchrony - Detection, pathophysiology, and clinical relevance: A Narrative review. Ann Thorac Med. 2020 Oct-Dec;15(4):190-198. doi: 10.4103/atm.ATM_63_20. Epub 2020 Oct 10. PMID 33381233
- [Result] Bachmann MC, Morais C, Bugedo G, Bruhn A, Morales A, Borges JB, Costa E, Retamal J. Electrical impedance tomography in acute respiratory distress syndrome. Crit Care. 2018 Oct 25;22(1):263. doi: 10.1186/s13054-018-2195-6. PMID 30360753